CLINICAL TRIAL: NCT04029675
Title: The Effect of High Dose of Vitamin C on the Clinical Outcome of Mechanically Ventilated Patients Following Sepsis in Intensive Care Unit
Brief Title: High Dose of Vitamin C on Mechanically Ventilated Septic Patients in Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Wessam Adel El Sayed Abdel Aziz El Driny, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Faculty of Pharmacy_AinShamsU
Record Dates: First submitted 2019-07-11; First posted 2019-07-23 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Ventilator Associated Pneumonia ( VAP); Sepsis
Keywords: Vitamin C; Sepsis; Intensive care unit; Mechanically ventilation; VAP
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Sepsis | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Double blinded ,Prospective, Randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group ( High dose vitamin C group ) (Experimental): They will receive 1.5 gm intravenous (IV) Vitamin C in 100 ml dextrose 5% (D5W) administered as an infusion over 30 to 60 minutes every 6 hours daily for 4 days or until ICU discharge.
  Interventions: Dietary Supplement: Vitamin C
- Control Group (Daily requirements vitamin C Group ) (Active Comparator): They will receive standard daily requirements of Vitamin C intravenously which is 75-90 mg in 100 ml dextrose 5% (D5W) administered as an infusion over 30 to 60 minutes daily for 4 days or until ICU discharge
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: Vitamin C — Vitamin C is a strong antioxidant and has been shown to regenerate other antioxidants such as vitamin E, vitamin C also play an important role in immune function

SUMMARY:
Prospective, Randomized clinical trial study will be carried out in intensive care unit in Ain Shams University Hospitals on 40 forty septic patients admitted to ICU and mechanically ventilated.

DETAILED DESCRIPTION:
This study will be carried out in intensive care unit in Ain Shams University Hospitals , Cairo,Egypt on 40 patients admitted to ICU that are septic patients and mechanically ventilated which will be recruited into the study . After approval from ethical committee, an informed consent will be obtained from relatives of all patients. All data of patients will be confidential with secret codes and private file for each patient. Each patient's relative will receive an explanation for the purpose of the study. The study design will be prospective , randomized clinical trial.

Methodology:

All patients will be subjected to:

1. Complete history taking.
2. Full clinical examination
3. Evaluation and monitoring of(pulse oximetry , ECG, NIBP, temperature)
4. CBC , Blood gas (for determination of (PaO2/FiO2), Blood cultures,serum Creatinine and total bilirubin were recorded daily for the first 7 days.
5. Severity scores by calculating Acute physiology and chronic health evaluation (APACHE II)score

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age from age≥18 years
* Septic patient admitted to ICU and mechanically ventilated diagnosed by sepsis criteria proposed by the American College of Chest Physicians/Society of Critical Care Medicine
* Expected to survive and remain in the ICU for at least 96 hours after study entry

Exclusion Criteria:

* Age<18 years
* Pregnant females
* Patients with history of aspiration before intubation
* Respiratory distress syndrome
* Ischemic reperfusion injury
* Cancer as the cause of SIRS or sepsis
* Chronic kidney diseases
* Ongoing shock
* Allergy from interventional drug on the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
The Incidence of Ventilator -Associated Pneumonia ( VAP) | within 28 days
  Ventilator-associated pneumonia (VAP)is defined as pneumonia that occurs 48-72 hours or thereafter following endotracheal intubation, characterized by the presence of a new progressive infiltrate, signs of a systemic infection (fever, altered white blood cells count), changes in sputum characteristics, and detection of a causative agent
Plasma Vitamin C level after administration of study drug | within 7 days of administered of vitamin C
  Vitamin C is a strong antioxidant and has been shown to regenerate other antioxidants such as vitamin E, vitamin C also play an important role in immune function
change in SOFA score | within 7 days of administered of vitamin C
  SOFA (Sepsis -related Organ Failure assessment) score

SECONDARY OUTCOMES:
28 day Mortality rate | average 28 days
length of stay in intensive care unit | through the study completion, average 6 months
changes in Glutathione Peroxidase enzyme (GPX) activity | within 7 days of administered of vitamin C
duration of vasopressor support | Average28 days
Ventilator-free days (28-days Cumulative ) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Sara M. Shahen, MD, Study Chair — Ain Shams University; Ibrahim E. Mamdoh, MD, Study Chair — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, EL Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No
data that to be shared are age & gender of the participants

REFERENCES:
- [Background] Annane D, Aegerter P, Jars-Guincestre MC, Guidet B; CUB-Rea Network. Current epidemiology of septic shock: the CUB-Rea Network. Am J Respir Crit Care Med. 2003 Jul 15;168(2):165-72. doi: 10.1164/rccm.2201087. PMID 12851245
- [Background] Martin GS, Mannino DM, Eaton S, Moss M. The epidemiology of sepsis in the United States from 1979 through 2000. N Engl J Med. 2003 Apr 17;348(16):1546-54. doi: 10.1056/NEJMoa022139. PMID 12700374
- [Background] Sands KE, Bates DW, Lanken PN, Graman PS, Hibberd PL, Kahn KL, Parsonnet J, Panzer R, Orav EJ, Snydman DR, Black E, Schwartz JS, Moore R, Johnson BL Jr, Platt R; Academic Medical Center Consortium Sepsis Project Working Group. Epidemiology of sepsis syndrome in 8 academic medical centers. JAMA. 1997 Jul 16;278(3):234-40. PMID 9218672
- [Background] Tanriover MD, Guven GS, Sen D, Unal S, Uzun O. Epidemiology and outcome of sepsis in a tertiary-care hospital in a developing country. Epidemiol Infect. 2006 Apr;134(2):315-22. doi: 10.1017/S0950268805004978. PMID 16490136
- [Background] Gogos CA, Drosou E, Bassaris HP, Skoutelis A. Pro- versus anti-inflammatory cytokine profile in patients with severe sepsis: a marker for prognosis and future therapeutic options. J Infect Dis. 2000 Jan;181(1):176-80. doi: 10.1086/315214. PMID 10608764
- [Background] CavaillonJ-M.Pathophysiological role of pro-and anti-inflammatory cytokines in sepsis .Sepsis.1998;2(2):127-40.
- [Background] Kurt AN, Aygun AD, Godekmerdan A, Kurt A, Dogan Y, Yilmaz E. Serum IL-1beta, IL-6, IL-8, and TNF-alpha levels in early diagnosis and management of neonatal sepsis. Mediators Inflamm. 2007;2007:31397. doi: 10.1155/2007/31397. PMID 18274637
- [Background] Oda S, Hirasawa H, Shiga H, Nakanishi K, Matsuda K, Nakamua M. Sequential measurement of IL-6 blood levels in patients with systemic inflammatory response syndrome (SIRS)/sepsis. Cytokine. 2005 Feb 21;29(4):169-75. doi: 10.1016/j.cyto.2004.10.010. Epub 2004 Dec 8. PMID 15652449
- [Background] Manzanares W, Biestro A, Torre MH, Galusso F, Facchin G, Hardy G. High-dose selenium reduces ventilator-associated pneumonia and illness severity in critically ill patients with systemic inflammation. Intensive Care Med. 2011 Jul;37(7):1120-7. doi: 10.1007/s00134-011-2212-6. Epub 2011 Mar 29. PMID 21445641
- [Background] Grossman RF, Fein A. Evidence-based assessment of diagnostic tests for ventilator-associated pneumonia. Executive summary. Chest. 2000 Apr;117(4 Suppl 2):177S-181S. doi: 10.1378/chest.117.4_suppl_2.177s. No abstract available. PMID 10816031
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Cook DJ, Walter SD, Cook RJ, Griffith LE, Guyatt GH, Leasa D, Jaeschke RZ, Brun-Buisson C. Incidence of and risk factors for ventilator-associated pneumonia in critically ill patients. Ann Intern Med. 1998 Sep 15;129(6):433-40. doi: 10.7326/0003-4819-129-6-199809150-00002. PMID 9735080
- [Background] Leroy O, Sanders V, Girardie P, Devos P, Yazdanpanah Y, Georges H, Beaucaire G. Mortality due to ventilator-associated pneumonia: impact of medical versus surgical ICU admittance status. J Crit Care. 2001 Sep;16(3):90-7. doi: 10.1053/jcrc.2001.28192. PMID 11689764
- [Background] Tejerina E, Frutos-Vivar F, Restrepo MI, Anzueto A, Abroug F, Palizas F, Gonzalez M, D'Empaire G, Apezteguia C, Esteban A; Internacional Mechanical Ventilation Study Group. Incidence, risk factors, and outcome of ventilator-associated pneumonia. J Crit Care. 2006 Mar;21(1):56-65. doi: 10.1016/j.jcrc.2005.08.005. PMID 16616625
- [Background] Visser J, Labadarios D, Blaauw R. Micronutrient supplementation for critically ill adults: a systematic review and meta-analysis. Nutrition. 2011 Jul-Aug;27(7-8):745-58. doi: 10.1016/j.nut.2010.12.009. PMID 21679878
- [Background] Sorice A, Guerriero E, Capone F, Colonna G, Castello G, Costantini S. Ascorbic acid: its role in immune system and chronic inflammation diseases. Mini Rev Med Chem. 2014 May;14(5):444-52. doi: 10.2174/1389557514666140428112602. PMID 24766384
- [Background] Fowler AA 3rd, Syed AA, Knowlson S, Sculthorpe R, Farthing D, DeWilde C, Farthing CA, Larus TL, Martin E, Brophy DF, Gupta S; Medical Respiratory Intensive Care Unit Nursing; Fisher BJ, Natarajan R. Phase I safety trial of intravenous ascorbic acid in patients with severe sepsis. J Transl Med. 2014 Jan 31;12:32. doi: 10.1186/1479-5876-12-32. PMID 24484547
- [Background] Tanaka H, Matsuda T, Miyagantani Y, Yukioka T, Matsuda H, Shimazaki S. Reduction of resuscitation fluid volumes in severely burned patients using ascorbic acid administration: a randomized, prospective study. Arch Surg. 2000 Mar;135(3):326-31. doi: 10.1001/archsurg.135.3.326. PMID 10722036
- [Background] Long CL, Maull KI, Krishnan RS, Laws HL, Geiger JW, Borghesi L, Franks W, Lawson TC, Sauberlich HE. Ascorbic acid dynamics in the seriously ill and injured. J Surg Res. 2003 Feb;109(2):144-8. doi: 10.1016/s0022-4804(02)00083-5. PMID 12643856
- [Background] - de GroothHJ,ChooWP,Spoelstra-deMan AMetal.Pharmacokinetics off our high- dose regimens of intravenousVitamin C in critically ill patients[Abstract]. IntensiveCareMed2016
- [Background] Padayatty SJ, Sun H, Wang Y, Riordan HD, Hewitt SM, Katz A, Wesley RA, Levine M. Vitamin C pharmacokinetics: implications for oral and intravenous use. Ann Intern Med. 2004 Apr 6;140(7):533-7. doi: 10.7326/0003-4819-140-7-200404060-00010. PMID 15068981
- [Background] Nathens AB, Neff MJ, Jurkovich GJ, Klotz P, Farver K, Ruzinski JT, Radella F, Garcia I, Maier RV. Randomized, prospective trial of antioxidant supplementation in critically ill surgical patients. Ann Surg. 2002 Dec;236(6):814-22. doi: 10.1097/00000658-200212000-00014. PMID 12454520
- [Background] Zabet MH, Mohammadi M, Ramezani M, Khalili H. Effect of high-dose Ascorbic acid on vasopressor's requirement in septic shock. J Res Pharm Pract. 2016 Apr-Jun;5(2):94-100. doi: 10.4103/2279-042X.179569. PMID 27162802
- [Background] Ascorbic Acid Injection.TheTorranceCompany,2015.
- [Background] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Result] Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Crit Care Med. 2001 Jul;29(7):1303-10. doi: 10.1097/00003246-200107000-00002. PMID 11445675
- [Derived] El Driny WA, Esmat IM, Shaheen SM, Sabri NA. Efficacy of High-Dose Vitamin C Infusion on Outcomes in Sepsis Requiring Mechanical Ventilation: A Double-Blind Randomized Controlled Trial. Anesthesiol Res Pract. 2022 Jul 15;2022:4057215. doi: 10.1155/2022/4057215. eCollection 2022. PMID 35873893